CLINICAL TRIAL: NCT04745117
Title: The Degree of Health Technologies Readiness Amongst Patients With Suspected Breast Cancer Using the READHY-tool
Brief Title: Health Technologies Readiness in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sollie, Medical doctor, Odense University Hospital
Other Study IDs: 21/4657
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Health Technology Readiness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with suspected breast cancer: All women referred under the diagnosis "suspected breast cancer" will be asked to fill out the questionnaire "READHY".
  Interventions: Behavioral: READHY - questionnaire

INTERVENTIONS:
Behavioral: READHY - questionnaire — The READHY tool consists of 70 questions divided into three sections, one with a focus on eHealth literacy, one on self-management and one on the social context. The READHY consists of the eHealth Literacy Questionnaire (eHLQ) that includes seven scales, supplemented with four scales from the Health Education Impact Questionnaire (heiQ) and two scales from the Health Literacy Questionnaire (HLQ). The READHY tool has been validated. Each question presented to the participant as a statement and scored on a 4-point rating, from 1=strongly disagree to 4=strongly agree. The overall score of each scale was calculated as the mean score of the 4-6 items (i.e., statements) that constitute the scale (2).

SUMMARY:
This study aims to investigate the degree of Health Technologies Readiness amongst patients with suspected breast cancer using the READHY-tool.

DETAILED DESCRIPTION:
Health information, patient education, and self-management (health information and advice) tools are increasingly being made available to adults with different health conditions, either through internet-based health and mobile health digital information technologies (1). At the department of plastic surgery, there has, for several years, been a transition to digital solutions when delivering information to patients. Patient information now consists of web-sites, apps and videos available for the patients to use when they seek information about their disease and their treatment options. From a care-givers perspective, the increased amount of information available is positive, but can these patients cope with so much information being available digitally instead of information face-to-face or by paper? Despite the rapid change from analogue informatics to digital solutions, we do not know a lot about our patients' readiness for such a change. There is an increasing amount of studies on the subject, but no recent study on readiness for digital solutions among this patient group, patients with suspected breast cancer. That is what this study is hoping to achieve with this study. The plan is to use a relatively new tool called "READHY" to assess the health technology readiness amongst breast cancer patients. The tool consists of 70 questions, and the results will enable grouping of these patients according to their health technology readiness.

This study is a cross-sectional study where participants fill out a single questionnaire at first contact with the out-patient clinic. There will not be any follow-up.

The project is planned to start at 01.03.2021 and run for six months with termination at 30.09.21.

A clinical statistician was consulted regarding power and sample size. No power analysis was performed due to the nature of the study. In accordance with previous studies with similar methods, a convenience sample was chosen. 250 participants will be included over six consecutive months (2,3).

All patient-reported data will be handled through the secure server solution provided by OPEN Region of Southern Denmark. Additional data will be kept in the secure server Sharepoint, provided by Odense University Hospital.

The project complies with The General Data Protection Regulation act (databeskyttelsesforordningen) and the Danish Data Protection act (databeskyttelsesloven).

The study is in line with the Helsinki-declaration. Participation is by individuals capable of giving informed consent.

There are no personal gains for our participants, but in the longer perspective, the information gathered will enable physicians to better understand the eHealth literacy in this patient group. This will, in turn, help to improve the way the patients arre informed about their disease, treatment and options.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to our department with suspected breast cancer.
* Ability to understand the aim of the study and to give consent. Being able to understand Danish at the level required to answer the questionnaires.

Exclusion Criteria:

* Danish skills that are insufficient for understanding and filling out the READHY-questionnaire in Danish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women referred to the Breast Cancer Center at Odense University Hospital under the suspicion of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Results of the Readiness and Enablement Index for Health Technology (READHY) | 1 month
  All participants will have a READHY-score calculated. Score ranges from 1-4. A higher score indicates a higher degree of health technology readiness.
Grouping using (Readiness and Enablement Index for Health Technology) READHY-scores | 6 months
  Using the results of the whole cohort, cluster analysis will be applied to group the participants into groups on levels of health technology readiness. Score ranges from 1-4. A higher score indicates a higher degree of health technology readiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No